CLINICAL TRIAL: NCT07023913
Title: Effect of Kinetic Control Exercise on Shoulder Dysfunction Post Mastectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Tarek Mostafa ElNawawy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alaa-005696
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Kinetic Control; Dysfunction; Shoulder; Mastectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinetic Control Exercise (Experimental): This group includes 30 patients who had mastectomy and will receive Kinetic control exercise inform of activation local and general Stabilizer, mobilizer), and traditional exercise. Patients will receive 3 sessions per week for 8 weeks.
  Interventions: Other: kinetic Control exercises; Other: traditional treatment
- traditional therapy (Active Comparator): This group includes 30 patients who have undergone mastectomy and will receive traditional therapy inform of stretching and strengthening exercise as shoulder roll, arm circle, wall climb, back climb and hand behind neck. Patients will receive 3 sessions per week for 8 weeks.
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: kinetic Control exercises — Kinetic Control exercises consist of 45-minute sessions, with 3 sessions per week for 8 weeks. The framework for testing and rehabilitation includes initial assessment, rehabilitation before failure, and retesting the same position. Biofeedback measures scapular retraction, and biofeedback pressure training assesses and improves scapular stabilizer control by monitoring pressure changes during specific movements.
  Arms: Kinetic Control Exercise
Other: traditional treatment — traditional therapy inform of stretching and strengthening exercise as shoulder roll, arm circle, wall climb, back climb and hand behind neck. Patients will receive 3 sessions per week for 8 weeks, the time of session is 45 - 60 min according to patient ability

SUMMARY:
The purpose of this study is to evaluate the effect of kinetic control exercises on shoulder dysfunction in post-mastectomy.

DETAILED DESCRIPTION:
This study holds significant importance for clinical practice, patient care, and research.

* Clinical Practice: It provides a potential framework for physical therapists to design targeted and effective interventions for shoulder dysfunction in post-mastectomy patients.
* Patient Care: Improved rehabilitation outcomes can enhance patients' physical functionality, independence, and overall quality of life, addressing a critical gap in post-operative recovery.
* Research Advancement: By contributing to the limited body of literature on kinetic control in this context, the study can stimulate further research and innovation in rehabilitative care for breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age from 40 to 50 years.
* All patients have no diabetes or blood problems.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Age less than 40 or more 50 years.
* Diabetes mellitus.
* Subjects with lymphedema
* Subjects suffering from active malignant tumors.
* Subjects treated with skin graft.
* Subjects with Mental illness.
* Subjects with skin diseases
* Subjects with any previous cause for shoulder dysfunction

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 60 female patient who will undergo mastectomy and suffers from post shoulder dysfunction. Their age will range from 40 to 50.
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
assessment of change of range of motion | at baseline and after 8 weeks
  Patients will be seated with their affected limb relaxed, and their goniometer will measure their resting position and active range. They will measure shoulder abduction and flexion, which are rarely affected by day-to-day activities, and external shoulder rotation.

SECONDARY OUTCOMES:
assessment of ability to maintain controlled shoulder movements while stabilizing the scapular and shoulder | at baseline and after 8 weeks
  it is a series of tests to assess kinetic control, including shoulder flexion, scapular retraction, and isometric holds. The tests focus on maintaining consistent pressure, detecting compensatory patterns, and evaluating fatigue. The tests also include a scapular stabilization test and a shoulder flexion stability test, which measure muscle activation patterns and stability.
assessment of ability to maintain controlled shoulder movements while stabilizing the scapular and shoulder | at baseline and after 8 weeks
  The tests also include a scapular stabilization test and a shoulder flexion stability test, which measure muscle activation patterns and stability.

CONTACTS AND LOCATIONS:
Locations (1):
- learning hospitals Al Kaser Al Ayni hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No